CLINICAL TRIAL: NCT02879123
Title: Assessment of Patients' Early Neurological Clinical Recovery, 3 Months After Endovascular Treatment of an Acute Ischemic Stroke
Brief Title: Early Neurological Clinical Recovery, 3 Months After Endovascular Treatment of an Acute Ischemic Stroke
Acronym: AVC-endovasc
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBC_2015_19
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This trial aims at collecting standardized data concerning the early neurological clinical recovery of patients, 3 months after endovascular treatment of an acute ischemic stroke.

Although this outcome is a major issue of patients' prognosis, it is rarely collected at this stage of their follow-up.

DETAILED DESCRIPTION:
Stroke affects 1 patient every 4 minutes in France, with around 130,000 new patients each year. Early recanalisation is a major prognostic factor and the main therapeutic target in the acute phase of this disease. The recanalisation techniques currently developed are intravenous thrombolysis, intra-arterial thrombolysis and thrombectomy (or embolectomy). These therapies can be combined. Thrombectomy involves endovascular capture of the clot obstructing the intracranial artery.

Recent improvements in thrombectomy techniques have also contributed to the spread of this technique. Neurovascular units include endovascular treatment in their strategy for the early management of acute proximal occlusions of intracranial arteries in almost 1 in 3 cases. This approach is currently the subject of professional agreements. Mechanical thrombectomy has now been validated by studies showing a major reduction (-35%) in the disability associated with severe cerebral infarction and a reduction in mortality, with recanalisation rates ranging from 58 to 72%. This "recanalisation" criterion is of major importance because it largely determines the functional prognosis of patients following a cerebral infarction.

Patients are often followed up in the months following the operation by the neurology department that initially treated them, and in the first few weeks they may be admitted to follow-up care units. As a result, although the clinical outcome at 3 months is a major factor in patient prognosis, this information is rarely available. The aim of this study is to obtain standardised 3-month follow-up data for a large series of patients who have undergone endovascular treatment for stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke
* endovascular treatment

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing endovascular treatment for an acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-11-12 (Actual); Primary Completion 2030-11-12 (Estimated); Study Completion 2031-05-12 (Estimated)

PRIMARY OUTCOMES:
early neurological clinical recovery | 3 months after endovascular treatment of an acute ischemic stroke
  modified RANKIN score

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Blanc, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France